CLINICAL TRIAL: NCT06079723
Title: Analyzing the Patterns of Patient Engagement and Trends in Participation Observed in Medullary Thyroid Cancer Clinical Trials
Brief Title: A Detailed Look At What Patients Experience In Medullary Thyroid Cancer Clinical Study
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 73927347
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Medullary Thyroid Cancer
Keywords: Medullary Thyroid Cancer
MeSH Terms: conditions — Carcinoma, Medullary

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical studies, with a distinct emphasis on medullary thyroid cancer, play a pivotal role in evaluating the safety and effectiveness of novel treatments for this condition. These trials serve as essential tools to determine whether new medications surpass conventional therapies, providing substantial evidence to endorse their broader adoption.

The primary objective is to meticulously examine trial completion rates and voluntary withdrawals within this specific patient group. By actively participating in this observational study plays a critical role in pushing medical knowledge forward and advancing care for individuals suffering from the medullary thyroid cancer.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of medullary thyroid cancer
* Aged ≥ 18 years old and ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed
* No serious medical or psychiatric illness likely to interfere with participation in this clinical study.

Exclusion Criteria:

* Is pregnant, breastfeeding or expecting to conceive within the projected duration of the study
* Any serious and/or unstable pre-existing medical disorders
* Patients who are currently receiving any other investigational drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Medullary thyroid cancer patients who are actively considering enrolling in an observational clinical study for said condition, but have not yet completed enrollment and randomization phases.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Number of medullary thyroid cancer patients who decide to enroll in a clinical trial | 3 months
Rate of medullary thyroid cancer patients who remain in clinical trial to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lam ET, Ringel MD, Kloos RT, Prior TW, Knopp MV, Liang J, Sammet S, Hall NC, Wakely PE Jr, Vasko VV, Saji M, Snyder PJ, Wei L, Arbogast D, Collamore M, Wright JJ, Moley JF, Villalona-Calero MA, Shah MH. Phase II clinical trial of sorafenib in metastatic medullary thyroid cancer. J Clin Oncol. 2010 May 10;28(14):2323-30. doi: 10.1200/JCO.2009.25.0068. Epub 2010 Apr 5. PMID 20368568
- [Background] Elisei R, Schlumberger MJ, Muller SP, Schoffski P, Brose MS, Shah MH, Licitra L, Jarzab B, Medvedev V, Kreissl MC, Niederle B, Cohen EE, Wirth LJ, Ali H, Hessel C, Yaron Y, Ball D, Nelkin B, Sherman SI. Cabozantinib in progressive medullary thyroid cancer. J Clin Oncol. 2013 Oct 10;31(29):3639-46. doi: 10.1200/JCO.2012.48.4659. Epub 2013 Sep 3. PMID 24002501
- [Background] Wells SA Jr, Robinson BG, Gagel RF, Dralle H, Fagin JA, Santoro M, Baudin E, Elisei R, Jarzab B, Vasselli JR, Read J, Langmuir P, Ryan AJ, Schlumberger MJ. Vandetanib in patients with locally advanced or metastatic medullary thyroid cancer: a randomized, double-blind phase III trial. J Clin Oncol. 2012 Jan 10;30(2):134-41. doi: 10.1200/JCO.2011.35.5040. Epub 2011 Oct 24. PMID 22025146

DOCUMENTS (1):
  • Informed Consent Form (2023-10-06): https://cdn.clinicaltrials.gov/large-docs/23/NCT06079723/ICF_000.pdf